CLINICAL TRIAL: NCT03232125
Title: Effect of Ramosetron on Heart Rate-corrected QT Interval During Robot-assisted Laparoscopic Prostatectomy With Steep Trendelenburg Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2017-0487
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ramosetron; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomly selected patients of the ramoseton group are given a 0.3 mg of ramosetron after induction. In contrast, patients in the control group are given the same volume of normal saline after induction and given a 0.3 mg of ramosetron after measurement of QTc interval.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, care provider and investigator are blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ramosetron group (Experimental): Randomly selected patients of the ramoseton group are given a 0.3 mg of ramosetron after induction.
  Interventions: Drug: Ramosetron
- Placebo group (Placebo Comparator): In contrast, patients in the control group are given the same volume of normal saline after induction and given a 0.3 mg of ramosetron after measurement of QTc interval.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ramosetron — Randomly selected patients of the ramoseton group are given a 0.3 mg of ramosetron after induction.
  Arms: Ramosetron group
Drug: Normal saline — In contrast, patients in the control group are given the same volume of normal saline after induction and given a 0.3 mg of ramosetron after measurement of QTc interval.
  Arms: Placebo group

SUMMARY:
Intraperitoneal insufflation of carbon dioxide may affect the sympathetic activity that leads to changes in ventricular re-polarization. This in turn can result in changes of heart rate-corrected QT (QTc) interval. Ramosetron is a 5-hydroxytryptamine three receptor antagonist and widely used anti-emetics. However, QTc interval prolongation has been observed in a number of patients after administration of 5-HT3 receptor antagonists. The aim of this study is to evaluate the effects of ramosetron on QTc interval and possible cardiovascular adverse effects during robot-assisted laparoscopic prostatectomy with steep Trendelenburg position.

DETAILED DESCRIPTION:
Intraperitoneal insufflation of carbon dioxide may affect the sympathetic activity that leads to changes in ventricular re-polarization. This in turn can result in changes of heart rate-corrected QT (QTc) interval. Ramosetron is a 5-hydroxytryptamine three receptor antagonist and widely used anti-emetics. However, QTc interval prolongation has been observed in a number of patients after administration of 5-HT3 receptor antagonists. The aim of this study is to evaluate the effects of ramosetron on QTc interval and possible cardiovascular adverse effects during robot-assisted laparoscopic prostatectomy with steep Trendelenburg position. Fifty-six patients, aged more than 19 years, undergoing robot-assisted laparoscopic prostatectomy will be divided into ramosetron group (n=28) and control group (n=28). Randomly selected patients of the ramoseton group are given a 0.3 mg of ramosetron after induction. In contrast, patients in the control group are given the same volume of normal saline after induction and given a 0.3 mg of ramosetron after measurement of QTc interval. The primary endpoint is the difference in maximal change of QTc interval between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing robot-assisted laparoscopic prostatectomy
* Age more than 19 years

Exclusion Criteria:

* Preoperative electrocardiography (ECG) abnormalities, including a QTc interval of >500 ms, ventricular conduction abnormalities, or arrhythmias
* History of cardiac disease such as pacemaker insertion, unstable angina
* Use of antiarrhythmic agents or medications that are known to prolong the QTc interval
* Abnormal levels of preoperative serum electrolyte

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Maximum change of QTc interval | Before induction of anesthesia in the supine position (Baseline)
  Maximum change of QTc interval from continuous ECG monitoring in lead V5 were collected by using the LabChart software.
Maximum change of QTc interval | 10 minutes after tracheal intubation (Intu-10 min.)
  Maximum change of QTc interval from continuous ECG monitoring in lead V5 were collected by using the LabChart software.
Maximum change of QTc interval | immediately after steep Trendelenburg position with CO2 pneumoperitoneum (T-on)
  Maximum change of QTc interval from continuous ECG monitoring in lead V5 were collected by using the LabChart software.
Maximum change of QTc interval | 30 minutes after steep Trendelenburg position with CO2 pneumoperitoneum (T-30 min)
  Maximum change of QTc interval from continuous ECG monitoring in lead V5 were collected by using the LabChart software.
Maximum change of QTc interval | 60 minutes after steep Trendelenburg position with CO2 pneumoperitoneum (T-60 min)
  Maximum change of QTc interval from continuous ECG monitoring in lead V5 were collected by using the LabChart software.
Maximum change of QTc interval | 90 minutes after steep Trendelenburg position with CO2 pneumoperitoneum (T-90 min)
  Maximum change of QTc interval from continuous ECG monitoring in lead V5 were collected by using the LabChart software.
Maximum change of QTc interval | immediately after a supine position with CO2 desufflation (T-off)
  Maximum change of QTc interval from continuous ECG monitoring in lead V5 were collected by using the LabChart software.
Maximum change of QTc interval | at the end of surgery (Surgery end)
  Maximum change of QTc interval from continuous ECG monitoring in lead V5 were collected by using the LabChart software.

CONTACTS AND LOCATIONS:
Locations (1):
- Professor, Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim TK, Cho YJ, Lim CW, Min JJ, Choi EK, Hong DM, Jeon Y. Effect of ramosetron on QTc interval: a randomised controlled trial in patients undergoing off-pump coronary artery bypass surgery. BMC Anesthesiol. 2016 Aug 3;16(1):56. doi: 10.1186/s12871-016-0222-1. PMID 27488394
- [Result] Lee JH, Yoo EK, Song IK, Kim JT, Kim HS. Effect of ramosetron on the QT interval during sevoflurane anaesthesia in children: a prospective observational study. Eur J Anaesthesiol. 2015 May;32(5):330-5. doi: 10.1097/EJA.0000000000000200. PMID 25485883
- [Result] Kim SH, Lee SM, Kim YK, Park SY, Lee JH, Cho SH, Chai WS, Jin HC. Effects of prophylactic ramosetron and ondansetron on corrected QT interval during general anesthesia. J Clin Anesth. 2014 Nov;26(7):511-6. doi: 10.1016/j.jclinane.2014.02.011. Epub 2014 Oct 18. PMID 25439413